CLINICAL TRIAL: NCT03043209
Title: Genomic Sequencing in Patients With Hypertrophic Cardiomyopathy Undergoing Septal Myectomy
Brief Title: Genomic Sequencing in Patients With HCM Undergoing Septal Myectomy
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Milind Desai, Medical Doctor, The Cleveland Clinic
Other Study IDs: 17-090
Record Dates: First submitted 2017-02-02; First posted 2017-02-03 (Estimated); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Hypertrophic Cardiomyopathy; Genetic Disease; Gene Product Sequence Variation
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — leftover of myectomy tissue and peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Genomic sequencing: Perform Genomic sequencing in peripheral blood DNA and discarded myocardium from cardiac procedures
  Interventions: Genetic: Genomic sequencing

INTERVENTIONS:
Genetic: Genomic sequencing — Genomic sequencing of DNA in Blood sample and myectomy tissue

SUMMARY:
Investigators aim to use comparative exome and/or genome sequencing to discover causative molecular lesions for phenotypes hypothesized to be caused by somatic mutations. For this study, investigators have targeted hypertrophic cardiomyopathy.

DETAILED DESCRIPTION:
The hypothesis is that sporadic or simplex occurrences of what are typically autosomal dominantly inherited diseases can instead be caused my mosaic mutations, specifically, mutations in the heart itself.

This hypothesis mandates that investigators sequence both affected and unaffected tissues, which in this case, investigators will construe to be peripheral blood DNA and discarded myocardium from cardiac procedures.

Eligible individuals will first undergo informed consent to be part of the study prior to their scheduled myomectomy. The study participants will also have phlebotomy for research samples.

The NIH Intramural Sequencing Center (NISC) will perform paired exome or genome sequencing and we will first screen for germline mutations in known cardiomyopathy genes that meet ACMG standards of likely pathogenic or pathogenic.

Then, if this is negative, investigators will screen for sequence variants that are present in cardiac tissue but absent in the blood DNA. Investigators will also screen blood DNA for secondary findings in genes recommended for annotation and results return by the ACMG and sequence variants deemed clinically relevant in this gene set will be validated in a CLIA-certified laboratory and the results returned to that participant.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years and older has a clinical diagnosis of hypertrophic cardiomyopathy.
* Patient scheduled for clinically-indicated myomectomy.
* Patient has a negative family history of hypertrophic cardiomyopathy
* Patient is willing to receive results of secondary variant screen

Exclusion Criteria:

* Pregnant
* Inability to give informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years and older, scheduled for septal myectomy and no family history of HCM
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2020-12-04 (Actual); Study Completion 2022-12-28 (Actual)

PRIMARY OUTCOMES:
Genetic causes of HCM in patients without a strong family history of the condition | one year
  The investigators will use DNA testing technology called "genomic sequencing"

CONTACTS AND LOCATIONS:
Overall Officials: Milind Desai, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided